CLINICAL TRIAL: NCT05593731
Title: Evaluation of Local Delivered Platelet Rich Fibrin Versus Melatonin Gel on the Osseointegration of Dental Implant. A Randomized Controlled Clinical Trial
Brief Title: Platelet Rich Fibrin Versus Melatonin Around Dental Implants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Radwa Elsherif, lecturer of oral medicine, periodontology, oral diagnosis, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Misprotocol
Record Dates: First submitted 2022-10-12; First posted 2022-10-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Patients With Missing Teeth
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dental implants alone (Other): dental implants alone
  Interventions: Biological: dental implants with melatonin gel
- platelet rich fibrin (Active Comparator): dental implants with platelet rich fibrin membrane
  Interventions: Biological: dental implants with melatonin gel
- melatonin gel (Active Comparator): dental implants with melatonin gel around dental implants
  Interventions: Biological: dental implants with melatonin gel

INTERVENTIONS:
Biological: dental implants with melatonin gel — platelet rich fibrin membrane around dental implants
  Other Names: dental implants with platelet rich fibrin

SUMMARY:
Dental implant is a dental treatment that allow oral rehabilitation for partial and fully edentulous patients. Osteointegration is the factor that control success s or failure of dental implant that can be improved by addition of different adjunctive biological materials. Platelets Rich fibrin plays a significant role in tissue regeneration and wound healing. Melatonin is biological hormone that secreted from pineal gland and played an important role in human growth.

ELIGIBILITY:
Inclusion Criteria:

1. good oral hygiene participants,
2. free of any systemic diseases,
3. Patients' age ranged from 20 to 40 years old.
4. Patients who can complete surgery and the study protocol.
5. Partially edentulous patients in the posterior mandibular region (at least a single-mandibular edentulous area) with periodontal health.

Exclusion Criteria:

1. patients who had parafunctional habits,
2. current and former smokers, pregnant
3. lactating women
4. unmotivated patients
5. patients with psychological problems
6. patients who were not able to follow the treatment protocol -

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female as melatonin is sex prevalence
Enrollment: 30 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
gingival thickness | 6 months

SECONDARY OUTCOMES:
bone density | 6 months
marginal bone loss | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry at MUST, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No